## **Brief Title**

The Effects of Group Social Work Intervention on Children's Emotional Intelligence, Emotion Regulation Skills and Empathy Tendencies

NCT Number: To be assigned upon registration approval

This document is prepared for ClinicalTrias gov registration; the NCT number will be added following approval of the registration.

**DOCUMENT DATE** 

**05 December 2025** 

## **Informed Consent Form (For Child Participants)**

Dear Participant,

This research is part of the doctoral dissertation conducted by Merve Ozkul, a student in the Department of Social Work at Selçuk University's Health Sciences Institute, under the supervision of Prof. Dr. Serap DASBAS. The purpose of the current study is to determine the effects of an emotion-focused group social work intervention on the emotion regulation skills, emotional intelligence, and empathic tendencies of children in need of protection. For this purpose, we plan to conduct various activities and interviews within the scope of a 12-week group study. Participation in the research is entirely voluntary. If you feel uncomfortable during the study, you may discontinue the study. No audio/video recordings will be taken of you during the study. Your name will not be used, directly or indirectly, in any documents generated as a result of this research. Your responses will be kept completely confidential, and the information obtained will be used solely for scientific purposes within the scope of this research. You may request that the data obtained as a result of your participation be excluded from the study at any time. For more information about the research or to access the results, please contact Merve OZKUL.

I am participating in this study entirely voluntarily and understand that I can discontinue my participation at any time. I agree to the use of the information I provide in scientific publications.

Date:

Participant Name-Surname:

## **Researcher Name and Surname:**

Merve OZKUL Selçuk University 0507-822-1469